CLINICAL TRIAL: NCT02948335
Title: Interactions of Environmental and Human Microbial Communities in a Pediatric Oncology Hospital
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NVIROM
Record Dates: First submitted 2016-10-18; First posted 2016-10-28 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Infection
Keywords: Microbial communities; Hospital environment; Disinfection; Adenosine triphosphate measures; Bioburden
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Microorganisms that colonize hospital environments play an important role in the transmission of hospital acquired infections (HAI) and multi-drug resistant organisms. Previous studies examining microorganisms in the hospital environment have been limited by reliance on targeted culture-based methods resulting in potentially missed or unrecognized organisms. Evidence now suggests that using microbiome analysis offers an innovative strategy that may improve our understanding of HAI and how best to prevent them.

This pilot longitudinal observational study aims to characterize the taxonomic composition of microbial communities on environmental surfaces and people in these environments prior to and following the introduction of patients, caregiver, and hospital staff to newly constructed inpatient care areas at St. Jude Children's Research Hospital (SJCRH). This proposed study is uniquely characterized by evaluating the hospital environment of a pediatric immunocompromised oncology patient population that has not been studied in the past using advanced molecular techniques such as microbiome analysis.

PRIMARY OBJECTIVE:

* To describe the pattern of microbial communities of the hospital environment before, during and after patient occupancy of a newly constructed hospital space.

SECONDARY OBJECTIVES:

* To describe the similarity or difference of environment microbial communities to that of the humans occupying this environment in a newly occupied hospital space.
* To describe the pattern in environment microbial communities after each step of disinfection (manual cleaning with chemical disinfectant and Ultraviolet light disinfection machine) after patient discharge from the inpatient hospital environment.
* To evaluate the correlation between environmental Adenosine Triphosphate (ATP) measures and organism bioburden.

DETAILED DESCRIPTION:
Participants will be recruited from the patient population at SJCRH. Patients admitted to one of the protocol defined inpatient rooms in the Kay Research and Care Center (KRCC) will be enrolled on the study. Participating patients will be asked to provide stool, nasal swab, and skin swab samples while inpatient. Primary caregivers and the nurse assigned to the patient's room will also be asked to provide nasal and skin swabs while the patient remains inpatient. These samples will be used to characterize the human microbiome for comparison to the environmental microbiome.

ELIGIBILITY:
Patient Participant Inclusion Criteria:

* Patients scheduled to be admitted or admitted to SJCRH,
* Admitted to one of the protocol defined inpatient rooms in the KRCC building at SJCRH,
* Patient, parents or legal guardian willing and able to provide informed consent and comply with study requirements,
* When applicable, participant is willing to provide assent and comply with the study requirements.

Patient Participant Exclusion Criteria:

* Inability or unwillingness of participant or legal guardian/representative to give written informed consent.

Primary Caregiver Participant Inclusion Criteria

* Primary caregiver anticipated to provide care for patient while he or she is inpatient at St. Jude Children's Research Hospital,
* ≥ 18 years old,
* Able and willing to provide informed consent and comply with study requirements.

Primary Caregiver Participant Exclusion Criteria

* Inability or unwillingness of primary caregiver to give informed consent.
* Primary Nurse Participant Inclusion Criteria
* Nurse assigned to patient participant on the day of patient participant sample collection
* Willing to provide informed consent

Primary Nurse Participant Exclusion Criteria

* Inability or unwillingness to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients and their nursing staff and caregivers admitted to the Kay Research and Care Center inpatient unit.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2018-02-19 (Actual); Study Completion 2018-02-19 (Actual)

PRIMARY OUTCOMES:
Change in diversity index of environment microbial composition | Before participant admission to after participant discharge, which is up to 30 days
  Microbial flora colonizing a newly built hospital environment will be compared prior to participant inpatient admission to after inpatient hospital discharge. Microbiome diversity is a measure of the richness of microbial species present in the environmental sample. It is reported as diversity index.
Change in microbiome composition within the environment microbial composition | Before participant admission to after participant discharge, which is up to 30 days
  Microbial flora colonizing a newly built hospital environment will be compared prior to participant inpatient admission to after inpatient hospital discharge. Microbiome composition describes which bacteria are detected in a sample. It is reported as percentage of relative abundance of each taxa of bacteria.

CONTACTS AND LOCATIONS:
Overall Officials: Hana Hakim, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org